CLINICAL TRIAL: NCT02923310
Title: Evaluation of Two Types of PRP in Knee Osteoarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Joyce Maria Annichino Bizzacchi, Professor, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19466713.6.0000.5404
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Osteoarthrits G II and III (Experimental): Group of treatment
  Interventions: Biological: Platelets Rich Plasma; Biological: Leucocyte - Platelets Rich Plasma; Drug: Hialuronic Acid
- Osteoarthrits GIV (Experimental): Group of treatment
  Interventions: Biological: Platelets Rich Plasma; Biological: Leucocyte - Platelets Rich Plasma; Drug: Hialuronic Acid

INTERVENTIONS:
Biological: Platelets Rich Plasma
Biological: Leucocyte - Platelets Rich Plasma
Drug: Hialuronic Acid

SUMMARY:
OOsteoarthritis (OA) is a chronic joint disease characterized by progressive degeneration of cartilage and bone tissue, leading to the appearance of subchondral cysts, osteophyte formation and synovial inflammation. Although the causes of OA are still poorly understood, biomechanical stresses able to reach the articular cartilage and subchondral bone, biochemical changes in cartilage and synovial membrane, as well as genetic factors are important items in its pathogenesis. Although there is no cure for OA, treatment is directed to each individual patient, seeking to minimize pain, maintain or improve joint range of motion and limit disability. New therapies able to accelerate regeneration and tissue repair process are being discussed. The viscosupplementation with hyaluronic acid (HA) have been shown to be an effective and safe treatment alternative in the fight against knee OA, in addition to HA, worth highlighting the therapeutic effects of growth factors derived from autologous platelets. The platelet-rich plasma (PRP) appears as an autologous therapy, non-immunogenic, able to induce healing and repair of bone soft tissue. This study aims to evaluate the clinical efficacy, comparing treatment with PRP and the combination of HA and PRP in the treatment of knee OA. To this, 120 will be selected OA patients with mild, moderate and severe (Grade II, III and IV). Selected patients will be scheduled for the procedures and randomly assigned randomly. In PRP be determined concentrations of the growth factor PDGF, TGFb 1, VEGF, EGF, by the method Bio Plex®.\. Functional evaluations will be conducted through questionnaires (WOMAC and SF-36) as measures of function and quality of self-reported life. The walking and strength test will be performed before and during periods of 90.180 and 360 days after the first application. The main motivation for the development of this study is the lack of randomized, double-blind clinical studies in the literature, and also based on the favorable results researchers have obtained, both with the use of HA, as the use of PRP in accelerating the process scar, preventing the development of arthrosis above. Therefore, we believe that the PRP, with its growth factors associated with synthetic HA play a synergistic action that should be studied in detail, in order to establish an effective therapeutic approach in the treatment of patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

Patients with Osteoarthrits

Exclusion Criteria:

* diabetes, rheumatoid arthritis, axial deviation (varus> 10 degrees valgus> 10 degrees), blood disorders (coagulopathy and platelet changes), cardiovascular diseases, infections, immunosuppression, patients on anticoagulant therapy or antiplatelet use of nonsteroidal anti-inflammatory 5 days before blood collection, patients with hemoglobin concentrations <11 and platelet count <150,000 mm³.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Womac | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hemotherapy and Hematology Center, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No